CLINICAL TRIAL: NCT05277012
Title: A Phase 1, Open-label, Randomized, Single-dose, Three-treatment, Three-way Crossover Pharmacokinetic Study to Evaluate the Relative Bioavailability of Etrumadenant (AB928) Tablet and Capsule Formulations and Food Effect on the Pharmacokinetics of the Tablet Formulation in Healthy Adult Participants
Brief Title: A Study to Evaluate Pharmacokinetics (PK) of Etrumadenant Tablet and Capsule Formulations in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARC-23
Record Dates: First submitted 2022-01-31; First posted 2022-03-14 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants
Keywords: Etrumadenant; Healthy participants; Pharmacokinetics; AB928; Tablet; Capsule

STUDY DESIGN:
Intervention Model Description: The study participants will receive 3 treatments (Treatment A, B and C) sequentially during the Treatment Period 1, 2, and 3.
  Treatment A: etrumadenant capsule in fasted state Treatment B: etrumadenant tablet in fasted state Treatment C: etrumadenant tablet in fed state Each treatment will be separated by a washout period of 7 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment sequence ABC (Experimental): Participants will be sequentially administered with Treatment A, B then C (Treatment A: etrumadenant capsule in fasted state; Treatment B: etrumadenant tablet in fasted state; Treatment C: etrumadenant tablet in fed state). Each treatment will be separated by a washout period of 7 days.
  Interventions: Drug: Etrumadenant
- Treatment sequence BCA (Experimental): Participants will be sequentially administered with Treatment B, C then A. Each treatment will be separated by a washout period of 7 days.
  Interventions: Drug: Etrumadenant
- Treatment sequence CAB (Experimental): Participants will be sequentially administered with Treatment C, A then B. Each treatment will be separated by a washout period of 7 days.
  Interventions: Drug: Etrumadenant

INTERVENTIONS:
Drug: Etrumadenant — Etrumadenant capsule and tablet formulations
  Other Names: AB928

SUMMARY:
This study will compare the pharmacokinetics (PK) effect of single-dose etrumadenant tablet and capsule formulations in fasted conditions. The effect of food on single-dose PK of tablet formulation will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female (non-childbearing potential), 19-55 years of age, inclusive, at the screening visit.
* Body mass index (BMI) between 18.0 and 32.0 kilograms/m^2 inclusive, at screening.
* Healthy as determined by medical history, physical examination, vital signs, and ECG assessed at the screening visit.
* Clinical laboratory test results clinically acceptable at screening and check in.
* Non-smokers or ex-smokers [must have ceased smoking and stopped using nicotine containing products greater than (>) 3 months prior to the first dosing] based on participant self-reporting.
* Able to swallow multiple capsules or tablets.

Exclusion Criteria:

* Participants who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, rheumatological, dermatological, endocrine, connective tissue diseases or disorders, in the opinion of the PI or designee.
* Have a clinically relevant surgical history, in the opinion of the PI or designee.
* History of relevant atopy or hypersensitivity to etrumadenant or related compounds.
* History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing.
* History (within 3 months of screening visit) of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 g of alcohol [equivalent to approximately 8 oz of beer (5.5% alcohol); 1 oz of 45% alcohol; or 3.5 oz of wine (12% alcohol)] based on self-reporting.
* Have a significant infection or known inflammatory process upon screening or check in, in the opinion of the PI or designee.
* Have acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea, heartburn) at the time of screening or check in.
* Female participants of childbearing potential.
* Positive results for hepatitis B, C, HIV-1 or HIV-2.
* Clinically significant hypokalemia in the opinion of the PI or designee.
* Have been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 30 days prior to the first dosing.
* Donation of blood or significant blood loss within 56 days prior to the first dosing.
* Plasma donation within 7 days prior to the first dosing.
* Participation in another clinical study within 30 days prior to the first dosing.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Etrumadenant | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Treatment Period 1, 2 and 3
Area Under the Plasma Concentration-time Curve From 0 to Last Observed Non-zero Concentration [AUC(0-t)] of Etrumadenant | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Treatment Period 1, 2 and 3
Area Under the Plasma Concentration Time Curve From Time '0' Extrapolated to Infinity [AUC(0-inf)] of Etrumadenant | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Treatment Period 1, 2 and 3
Time to Cmax (Tmax) of Etrumadenant | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Treatment Period 1, 2 and 3
Apparent First-order Terminal Elimination Rate Constant (Kel) of Etrumadenant | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Treatment Period 1, 2 and 3
Percentage of AUC(0-inf) Extrapolation (AUC%extrap) of Etrumadenant | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Treatment Period 1, 2 and 3
Apparent First Order Terminal Elimination Half-life (t1/2) of Etrumadenant | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Treatment Period 1, 2 and 3
Apparent Total Plasma Clearance (CL/F) of Etrumadenant | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Treatment Period 1, 2 and 3
Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) of Etrumadenant | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Treatment Period 1, 2 and 3
Ratio of Etrumadenant metabolites to Etrumadenant | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Treatment Period 1, 2 and 3
Ratio of Etrumadenant metabolites to Total Metabolite Concentration | Multiple timepoint evaluations from pre-dose to 24 hours post-dose at Days 1, 2, 3, 4, 5, and 6 during Treatment Period 1, 2 and 3

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 4 months
  Safety will be assessed by monitoring adverse events and clinically significant changes in 12 lead Electrocardiogram, vital signs, and clinical laboratory tests results.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (1):
- Investigational Site, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy